CLINICAL TRIAL: NCT00653276
Title: An Open-Label, 2-Period, Crossover Study to Determine the Effect of Multiple Oral Doses of Ezetimibe 20 mg on the Pharmacokinetics of a Single Oral Dose of Cyclosporine in Young, Healthy, Normal, Male and Female Subjects
Brief Title: MD Ezetimibe Cyclosporine Interaction (0653-057)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0653-057; MK0653-057; 2008_520
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Cholesterol
MeSH Terms: interventions — Ezetimibe

ARMS (2):
- Treatment A (Active Comparator): Treatment A: subjects will be given a single oral dose of cyclosporine 100 mg capsules on Day 1.
  Interventions: Drug: Comparator: cyclosporine
- Treatment B (Active Comparator): Treatment B: subjects will receive single oral daily doses of ezetimibe 20 mg (2 x 10 mg tablets) on Days 1 through 6, followed by coadministration of a single oral dose of ezetimibe 20 mg (2 x 10 mg tablets) and cyclosporine 100 mg capsule on Day 7.
  Interventions: Drug: ezetimibe; Drug: Comparator: cyclosporine

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 20 mg (2 x 10 mg tablets) on Days 1 through Day 7.
  Other Names: MK0653; Zetia®
  Arms: Treatment B
Drug: Comparator: cyclosporine — single oral dose of cyclosporine 100 mg capsules on Day 1 or Day 7.

SUMMARY:
Study to determine the effect of multiple oral doses of ezetimibe on the pharmacokinetics of a single oral dose cyclosporine in young healthy males and females.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 18 to 45 years of age
* Subject is judged to be in good health on the basis of history, physical examination, and routine laboratory data

Exclusion Criteria:

* Premenopausal women who are currently pregnant or who are currently nursing
* Subjects with drug or substance abuse, poor mental function, history of major gastrointestinal abnormalities (stomach issues), or high cholesterol
* Subject that has donated blood or has participated in another clinical trial within the last four weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2003-11; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of cyclosporine coadministered with ezetimibe vs. cyclosporine administered alone. | Blood sampling will be conducted for 48 hours starting with the first cyclosporine dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bergman AJ, Burke J, Larson P, Johnson-Levonas AO, Reyderman L, Statkevich P, Kosoglou T, Greenberg HE, Kraft WK, Frick G, Murphy G, Gottesdiener K, Paolini JF. Effects of ezetimibe on cyclosporine pharmacokinetics in healthy subjects. J Clin Pharmacol. 2006 Mar;46(3):321-7. doi: 10.1177/0091270005284851. PMID 16490808